CLINICAL TRIAL: NCT05532995
Title: Kinetics of Physiological and Symptomatic Responses to CardioPulmonary Exercise Testing (CPET) in Subjects With Persistent Exercise Intolerance After COVID-19: an Open-Source Exercise Network
Brief Title: Responses to CPET in Subjects With Persistent Exercise Intolerance After COVID-19: an Open-Source Exercise Network
Status: Completed | Type: Observational
Sponsor: Association pour la Complementarite des Connaissances et des Pratiques de la Pneumologie (Other)
Collaborators: Menarini Group (Industry); Hylab, Grenoble (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ACCPP-PROT2022-01
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
Keywords: Long COVID; Exercise test; Post-acute COVID syndrome; Sars-Cov-2; Multi-centric study; Respiration; Dyspnoea; Exercise intolerance; Fatiguability; Open-Source Network
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Respiratory Aspiration; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective collaborative study on persistent exercise intolerance after COVID-19 offers to perform a large descriptive analysis of CPET performed in real-life by pulmonologists, cardiologists and physiologists. Indeed, these practicians are regularly consulted for a persistent intolerance to exercise expressed by dyspnea and/or frank fatigability sometimes associated with muscular or thoracic pain. When these complaints persist beyond 3 months after the first symptoms, it is legitimate to perform a CPET:

* Either to evaluate the functional impact of an identified organ deficiency (e.g. myocarditis, pulmonary fibrosis, etc.),
* Or, in the absence of formal arguments for an identified organ deficiency, to observe possible abnormalities in physiological responses during an incremental exercise test, likely to explain the persistence of symptoms and intolerance to exercise. Indeed, the recent literature highlights the presence of non-specific ventilatory and cardio-circulatory abnormalities leading to various physio-pathological observations. Unfortunately, these reports now concern relatively small numbers of patients with very diverse clinical forms of Covid, comorbidities and habitus.

In order to improve the understanding of persistent symptoms and in particular the diversity of physiological response presentations, the investigators propose to collect a very large amount of data through a web-based platform designed to collect the measurements made throughout the exercise test directly from the ergospirometer.

The relevant data covers the period from January 2, 2020 to December 31, 2022 (i.e. 35 months), The retrospective data collection will be carried out from February 1, 2023 to December 31, 2023.

The descriptive analysis will focus on the kinetics of all the variables measured and calculated on subgroups defined a priori on age, sex, comorbidities, acute covid severity, persistent symptoms post covid, regular habitual physical activity level, etc. according to the sample.

The study is expected to collect data from around 1000 patients and to involve around 40 French-speaking investigators. However, this collaborative study is open on request to all centers wishing to participate, as the web platform has been developed for data collection in English.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with persistent symptoms 3 months after the onset of Covid-19 infection, regardless the severity of the initial illness
* Patients with an ICU stay, primarily following rehabilitation management; that is, in practice, at least 6 months after COVID
* Patients followed by a pulmonologist, cardiologist or physiologist in a public or private facility or in private practice, allowing for CPET
* Patients who have performed a CPET before December 31, 2023
* Patients informed of the possible anonymized processing of the data collected during CPET for research purposes; and who gave informed consent

Exclusion Criteria:

* Age < 18 years
* Patients unable to perform CPET for locomotor reasons
* Patients with severely reduced functional work capacity
* Patient deprived of liberty by judicial or administrative decision
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with exercise intolerance after COVID-19, diagnosed between January 2, 2020 and December 31, 2023, who have been informed that the physiological data collected during the CPET and the clinical data necessary for its interpretation may be used for clinical research.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
An abnormal CPET due to either decreased respiratory capacity, excessive dyspneoa, deconditioning or breathing disorder | A descriptive analysis of all evaluation criteria will be performed on the total population and on subgroups to be defined a posteriori according to the sample (December 2023).

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Aguilaniu, M.D. PhD, Study Director — Association pour la Complementarite des Connaissances et des Pratiques de la Pneumologie; PierAntonio Laveneziana, M.D. PhD, Principal Investigator — University Hospital La Pitié-Salpêtrière; Frédéric Costes, M.D. PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (29):
- Hosp. Maisonneuve-Rosemont, Montreal, Canada
- France (26):
  - University Hosp. Amiens-Picardie, Amiens
  - Angers University Hosp., Angers
  - AP-HP University Hosp. Avicenne, Bobigny
  - Brest University Hosp. Cavale Blanche, Brest
  - Hosp. Louis Pradel, Bron
  - SSR Marguerite Boucicaut French Red Cross, Chalon-sur-Saône
  - University Hosp. Gabriel-Montpied, Clermont-Ferrand
  - Corbie General Hosp. (Réadaptation), Corbie
  - Centre de Réadaptation Cardio-Respiratoire Dieulefit Santé, Dieulefit
  - Centre Médical Bayère, Gleizé
  - Grenoble Alpes University Hosp. Michallon Nord, Grenoble
  - Grenoble Alpes University Hosp. Michallon Sud, Grenoble
  - Hosp. St Philibert GH Catholique Institute Lille, Lille
  - Limoges General Hosp., Limoges
  - Medical Center Parot, Lyon
  - Médipôle Lyon-Villeurbanne, Lyon
  - Nice University Hosp. Pasteur, Nice
  - Clinique Les Rieux, Nyons
  - AP-HP Hôpital Bichat Claude-Bernard, Paris
  - AP-HP University Hosp. Cochin, Paris
  - AP-HP University Hosp. Pitié Salpêtrière, Paris
  - Polyclinique Les Bleuets, Reims
  - University Hosp. of Pontchaillou, Rennes
  - Rouen University Hosp. Charles-Nicolle, Rouen
  - Toulouse University Hosp., Toulouse
  - Tours University Hosp. Bretonneau, Tours
- Clinique Saint Paul, Fort-de-France, Martinique
- Geneva University Hosp., Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gao Y, Chen R, Geng Q, Mo X, Zhan C, Jian W, Li S, Zheng J. Cardiopulmonary exercise testing might be helpful for interpretation of impaired pulmonary function in recovered COVID-19 patients. Eur Respir J. 2021 Jan 28;57(1):2004265. doi: 10.1183/13993003.04265-2020. Print 2021 Jan. PMID 33361097
- [Background] Cortes-Telles A, Lopez-Romero S, Figueroa-Hurtado E, Pou-Aguilar YN, Wong AW, Milne KM, Ryerson CJ, Guenette JA. Pulmonary function and functional capacity in COVID-19 survivors with persistent dyspnoea. Respir Physiol Neurobiol. 2021 Jun;288:103644. doi: 10.1016/j.resp.2021.103644. Epub 2021 Feb 27. PMID 33647535
- [Background] Gervasi SF, Pengue L, Damato L, Monti R, Pradella S, Pirronti T, Bartoloni A, Epifani F, Saggese A, Cuccaro F, Bianco M, Zeppilli P, Palmieri V. Is extensive cardiopulmonary screening useful in athletes with previous asymptomatic or mild SARS-CoV-2 infection? Br J Sports Med. 2021 Jan;55(1):54-61. doi: 10.1136/bjsports-2020-102789. Epub 2020 Oct 5. PMID 33020140
- [Background] Mohr A, Dannerbeck L, Lange TJ, Pfeifer M, Blaas S, Salzberger B, Hitzenbichler F, Koch M. Cardiopulmonary exercise pattern in patients with persistent dyspnoea after recovery from COVID-19. Multidiscip Respir Med. 2021 Jan 25;16(1):732. doi: 10.4081/mrm.2021.732. eCollection 2021 Jan 15. PMID 33623700
- [Background] Townsend L, Moloney D, Finucane C, McCarthy K, Bergin C, Bannan C, Kenny RA. Fatigue following COVID-19 infection is not associated with autonomic dysfunction. PLoS One. 2021 Feb 25;16(2):e0247280. doi: 10.1371/journal.pone.0247280. eCollection 2021. PMID 33630906
- [Background] Motiejunaite J, Balagny P, Arnoult F, Mangin L, Bancal C, d'Ortho MP, Frija-Masson J. Hyperventilation: A Possible Explanation for Long-Lasting Exercise Intolerance in Mild COVID-19 Survivors? Front Physiol. 2021 Jan 18;11:614590. doi: 10.3389/fphys.2020.614590. eCollection 2020. PMID 33536937
- [Background] Debeaumont D, Boujibar F, Ferrand-Devouge E, Artaud-Macari E, Tamion F, Gravier FE, Smondack P, Cuvelier A, Muir JF, Alexandre K, Bonnevie T. Cardiopulmonary Exercise Testing to Assess Persistent Symptoms at 6 Months in People With COVID-19 Who Survived Hospitalization: A Pilot Study. Phys Ther. 2021 Jun 1;101(6):pzab099. doi: 10.1093/ptj/pzab099. PMID 33735374
- [Background] Dorelli G, Braggio M, Gabbiani D, Busti F, Caminati M, Senna G, Girelli D, Laveneziana P, Ferrari M, Sartori G, Dalle Carbonare L, Crisafulli E, On Behalf Of The Respicovid Study Investigators. Importance of Cardiopulmonary Exercise Testing amongst Subjects Recovering from COVID-19. Diagnostics (Basel). 2021 Mar 12;11(3):507. doi: 10.3390/diagnostics11030507. PMID 33809260
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1qiU0UgEzvPBntfA0lLWFe_AzOGngacl9/view?usp=sharing

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT05532995/Prot_ICF_001.pdf